CLINICAL TRIAL: NCT00909792
Title: Clinical Evaluation of Two New Silicone Hydrogel Multifocal Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-319-C-013
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lotrafilcon B / Senofilcon A (Other): Lotrafilcon B, followed by Senofilcon A
  Interventions: Device: Lotrafilcon B; Device: Senofilcon A
- Senofilcon A / Lotrafilcon B (Other): Senofilcon A, followed by Lotrafilcon B
  Interventions: Device: Lotrafilcon B; Device: Senofilcon A

INTERVENTIONS:
Device: Lotrafilcon B — Silicone hydrogel, soft, multifocal contact lens
Device: Senofilcon A — Silicone hydrogel, soft, multifocal contact lens

SUMMARY:
The objective of this trial is compare the visual performance, ratings, and preference of two multifocal, soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 35 years of age
* Best-corrected distance visual acuity of at least 20/40 in each eye.
* Spectacle add between +0.75D and +1.50D (inclusive).
* Able to be fit in available study sphere powers (-1.00 to -5.00D)
* Currently wearing soft contact lenses at least 5 days a week.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* Astigmatism ≥ 1.00D.
* Currently wearing either of the study products.
* Other protocol inclusion/exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but not dispensed due to failing inclusion/exclusion criteria. This participant is included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Groups:
- Lotrafilcon B / Senofilcon A: Lotrafilcon B multifocal contact lenses worn first, with Senofilcon A multifocal contact lenses worn second. Both products worn in a daily wear basis.
- Senofilcon A / Lotrafilcon B: Senofilcon A multifocal contact lenses worn first, with Lotrafilcon B multifocal contact lenses worn second. Both products worn in a daily wear basis.
Period: Period 1
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 130 | 128
Completed | 130 | 127
Not Completed | 0 | 1
Not completed — Did not meet inclusion criteria | 0 | 1
Period: Period 2
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 129 (One participant discontinued between Period 1 and Period 2 due to lack of efficacy.) | 125 (Two discontinuations between P1 & P2: 1 for fail inc/exc criteria; 1 for lack of efficacy.)
Completed | 128 | 124
Not Completed | 1 | 1
Not completed — Biomicroscopy | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 258
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Binocular Visual Measurement in Normal Illumination Reported as Binocular Distance Visual Acuity
Description: Tested while reading charts distant to the subject with both eyes together in normal lighting. This outcome is measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 equates to 20/20 Snellen acuity and is considered normal. Positive logMAR values indicate poorer vision and negative values denote better visual acuity.
Time Frame: After 1 week of wear
Population: Per Protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Lotrafilcon B Multifocal Contact Lens; Senofilcon A Multifocal Contact Lens: Silicone hydrogel, soft, multifocal contact lens
Arm/Group | Lotrafilcon B Multifocal Contact Lens | Senofilcon A Multifocal Contact Lens
Number analyzed (Participants) | 237 | 234
logMAR | -0.01 (0.06) | 0.01 (0.07)

ADVERSE EVENTS:
Time Frame: 46 days, duration of the study.
Arm/Group | Lotrafilcon B | Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/256 | 0/258
Other Adverse Events (participants affected / at risk) | 0/256 | 0/258

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any pre-clinical and/or clinical data or impressions from this trial.